CLINICAL TRIAL: NCT00276926
Title: Open Label Pilot Phase II Study of STI571 in the Treatment of Patients With Idiopathic Hypereosinophilic Syndrome (HES) and Eosinophilic Leukemias
Brief Title: Study of STI571 in the Treatment of Patients With Idiopathic Hypereosinophilic Syndrome (HES) and Eosinophilic Leukemias
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HES0203
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Hypereosinophilic Syndrome; Chronic Eosinophilic Leukemia (CEL); Myeloproliferative Disorders
Keywords: Hypereosinophilic Syndrome; Eosinophilic leukemias; STI571 (Gleevec); PDGF receptor alpha; Familiar hypereosinophilia; Myeloproliferative disorder (MPD) with eosinophilia; myeloproliferative disorders/myelodysplastic syndromes
MeSH Terms: conditions — Hypereosinophilic Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: STI571

SUMMARY:
The purpose of this study is to assess the clinical anti-proliferative activity of STI571 (Glivec®, Novartis, Pharma) in patients with HES defined as:

1. Idiopathic Hypereosinophilic Syndrome (secondary HES), defined as a peripheral blood eosinophilia greater than 1,500 cells/µL for longer than 6 months, absence of other apparent aetiologies for eosinophilia and with or without signs and symptoms of organ involvement, irrespective to expression of any of imatinib targets (c-Kit receptor, PDGFR, bcr-abl receptor) on bone marrow cells.
2. Familiar hypereosinophilia defined as a peripheral blood eosinophilia greater than 1,500 cells/µL for longer than 6 months, absence of other apparent aetiologies for eosinophilia and signs and symptoms of organ involvement, irrespective to expression of any of imatinib targets (c-Kit receptor, PDGFR, bcr-abl receptor) on bone marrow cells, and with a recognized or reported cases of hypereosinophilia in the patient's family.
3. Chronic myeloproliferative disorder, defined as chronic eosinophilic leukemia (CEL) with the presence of blasts (>10%) in the bone marrow (BM), or the presence of immature eosinophils in different tissues, or an aggressive clinical course or the presence of clonal cytogenetic anomalies.
4. Myeloproliferative disorder (MPD) with eosinophilia, eosinophilic leukemia or chronic myelomonocytic leukemia [myeloproliferative disorders/myelodysplastic syndromes (MPD/MDS)] with evidence of:

   * t(5;12)(q33;p13) by cytogenetic or fluorescent in situ hybridization (FISH) analysis, or
   * ETV6/TEL-PDGFRB fusion transcript by reverse transcription polymerase chain reaction (RT-PCR), or
   * PDGFRB disruption, assessed or suspected, by other translocations with additional partner genes (H4, HIP1, CEV14 and Rab5) 5, or
   * MPD/MDS who have constitutive activation of the gene for platelet-derived growth factor receptor beta (PDGFRB) 6 by point mutations

ELIGIBILITY:
Inclusion Criteria:

1. Presence of primary or secondary HES
2. Not a candidate for allogeneic bone marrow transplantation.
3. ECOG performance score of 0, 1, 2 or 3 (Karnofsky performance score > 40%).
4. Life expectancy > 4 weeks.
5. Adequate hepatic and renal function, as defined by serum transaminases < 2.5x upper limits of normal (ULN), bilirubin < 1.5x ULN, and creatinine < 1.5x ULN.
6. Age 18 years or greater.
7. Post-menopausal, surgically sterile, or taking effective contraception in female patients.
8. Documentation of written informed consent to participate in the trial.
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

1. Patients with clear evidence of secondary hypereosinophilia.
2. Acute myeloblastic leukemia with inv(16) positive blast or
3. CBFb-MYH11 transcripts positive leukemia
4. Lack of recovery from the acute toxic effects of previous chemotherapy [to common toxicity criteria (CTC) grade > 1] with the exception of chemotherapy-induced alopecia.
5. Treatment with any investigational agent within 4 weeks prior to study therapy.
6. Major surgeries within 4 weeks from study start or not fully recovered from any previous surgical procedure.
7. Presence of any medical or psychiatric condition which may limit full compliance with the study or increase the risk associated with study participation or study drug administration, including but not limited to
8. Presence of central nervous system (CNS) illness and involvement of disease.
9. Active uncontrolled bacterial infection.
10. Known human immunodeficiency virus (HIV) infection.
11. Grade 3 or 4 bleeding.
12. Significant cardiovascular disease (i.e., uncontrolled arrhythmias, unstable angina), or a major thromboembolic event (myocardial infarction, stroke, transient ischemic attack, pulmonary embolism, or non-catheter-related deep-vein thrombosis) in the last 6 months. Due to the low cardiac toxicity profile of Glivec, it is not considered an exclusion criterion if the presence of severe complications to the viscera, among which cardiopathies, and in particular endomyocardial fibrosis, is due or considered to be due to HES.
13. Increased blood eosinophil counts due to the presence of physician-diagnosed asthma. However, due to low pulmonary toxicity profile of Glivec, it is not considered an exclusion criterion, if HES is associated with asthma, and the presence of severe complications damaging the lungs, are considered due to HES.
14. Pregnancy or breast-feeding.
15. Malabsorption syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03

PRIMARY OUTCOMES:
Rate of complete response (CR) in all patients at 3rd month

SECONDARY OUTCOMES:
Duration of response (CR)
Overall survival at 12th month

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli" Università degli Studi di Bologna
Locations (14):
- Italy (14):
  - Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli" Università degli Studi di Bologna, Bologna
  - Dipartimento di Medicina Interna - Università di Genova, Genova
  - Dipartimento di Biochimica e Biotecnologie Mediche - Università degli Studi di Napoli "Federico II", Napoli
  - Divisione di Ematologia - Università degli Studi di Napoli "Federico II", Napoli
  - S.C. Medicina Interna II ed Ematologia - Laboratorio di Medicina Interna e Molecolare - A.O. San Luigi, Orbassano
  - Divisione di Ematologia - IRCCS Policlinico S. Matteo, Pavia
  - U.O. Ematologia - Dipartimento di Oncologia ed Ematologia, Presidio Ospedaliero di Ravenna, Ravenna
  - U.O. Ematologia - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Cattedra di Ematologia - Università "Tor Vergata", Roma
  - Cattedra di Ematologia - Università "La Sapienza", Roma
  - Divisione di Ematologia - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - Policlinico "Le Scotte", Siena
  - U.O. Medicina II Divisione - Ospedale Santa Chiara, Trento
  - Clinica Ematologica - Policlinico Universitario, Udine